CLINICAL TRIAL: NCT01404572
Title: Randomized, Double Blind, Crossover Taste Assessment Study of Two Atazanavir Powder Formulations As Compared to a Reference Atazanavir Powder Formulation in Healthy Subjects
Brief Title: Taste Assessment Study of 2 Atazanavir Powder Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: AI424-466
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-05

CONDITIONS: HIV
MeSH Terms: interventions — Atazanavir Sulfate; Powders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Atazanavir + 10% aspartame (Active Comparator)
  Interventions: Drug: Atazanavir (current formulation)
- Atazanavir + 4.2% aspartame (Active Comparator)
  Interventions: Drug: Atazanavir, powder for oral use 1 (POU1)
- Atazanavir + 4.2% aspartame and sucralose (Active Comparator)
  Interventions: Drug: Atazanavir (POU2)

INTERVENTIONS:
Drug: Atazanavir (current formulation) — Solution, oral, atazanavir 15 mg/5 mL with 10% aspartame, single dose
  Other Names: Reyataz
  Arms: Atazanavir + 10% aspartame
Drug: Atazanavir, powder for oral use 1 (POU1) — Solution, oral, atazanavir 15 mg/5 mL with 4.2% aspartame, single dose
  Other Names: Reyataz
  Arms: Atazanavir + 4.2% aspartame
Drug: Atazanavir (POU2) — Solution, oral, atazanavir 15 mg/5 mL with 4.2% aspartame and sucralose, single dose
  Other Names: Reyataz
  Arms: Atazanavir + 4.2% aspartame and sucralose

SUMMARY:
The purpose of this study is to compare the sweetness of 2 new atazanavir powder for oral use (POU) formulations to the current atazanavir POU in healthy participants and to select 1 atazanavir POU that has the sweetness most similar to the current atazanavir POU.

DETAILED DESCRIPTION:
This study is a taste assessment study designed to select a new atazanavir powder for oral use (POU) formulation that is similar in sweetness to the current POU formulation. Participants were to taste and then spit out the POU formulations, without swallowing them. Study Classification: Other. This is a taste study

ELIGIBILITY:
Key inclusion criteria:

* Healthy men and women, ages 18 to 49, inclusive
* Nonsmokers
* Women not pregnant or breastfeeding
* Participants who could match solutions of the same sweetness and provide consistent sweetness scores during the taste screening

Key exclusion criteria:

* Any significant acute or chronic medical illness
* Any acute or chronic condition that may have altered taste sensory perception
* Any major surgery or trauma within 4 weeks of Day 1
* Blood transfusion within 4 weeks of study participation
* Recent (within 6 months of Day 1) drug or alcohol abuse as defined in the Diagnostic and Statistical Manual, 4th edition, Diagnostic Criteria for Drug and Alcohol Abuse
* Positive urine drug screen
* Positive urine screen for cotinine
* Positive hepatitis C antibody, hepatitis B surface antigen, or human immunodeficiency virus antibodies
* Clinically significant elevations in results of liver function tests above normal range

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Pra International, Lenexa, Kansas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 12 participants were enrolled in this study, and all 12 received study drug within each treatment sequence.
Groups:
- Treatment Sequence A, B, C: Participants in this sequence first tasted (Treatment A) atazanavir, 15 mg/5 mL, powder for oral use (POU) in the current formulation with 10% aspartame followed by at least a 45-minute washout period. Next, participants tasted (Treatment B) atazanavir, 15 mg/5 mL, in the first new POU (POU1) with 4.2% aspartame. Following another at least 45-minute washout period, participants tasted (Treatment C) atazanavir, 15 mg/5 mL, in the second new POU formulation (POU2) with 4.2% aspartame plus 0.53% sucralose.
- Treatment Sequence B, C, A: Participants in this sequence first tasted (Treatment B) atazanavir, 15 mg/5 mL, in the first new POU (POU1) with 4.2% aspartame. Following at least a 45-minute washout period, participants tasted (Treatment C) atazanavir, 15 mg/5 mL, in the second new POU formulation (POU2) with 4.2% aspartame plus 0.53% sucralose. Following another 45-minute washout period, participants then tasted (Treatment A) atazanavir, 15 mg/5 mL, powder for oral use (POU) in the current formulation with 10% aspartame.
- Treatment Sequence C, A, B: Participants in this sequence first tasted (Treatment C) atazanavir, 15 mg/5 mL, in the second new POU formulation (POU2) with 4.2% aspartame plus 0.53% sucralose followed by at least a 45-minute washout period. Next, participants tasted (Treatment A) atazanavir, 15 mg/5 mL, powder for oral use (POU) in the current formulation with 10% aspartame. Following another at least 45-minute washout period, participants tasted (Treatment B) atazanavir, 15 mg/5 mL, in the first new POU (POU1) with 4.2% aspartame.
Period: Overall Study
Arm/Group | Treatment Sequence A, B, C | Treatment Sequence B, C, A | Treatment Sequence C, A, B
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Treated: All participants tasted atazanavir, 15 mg/5 mL, in the current formulation and 2 new powder for oral use formulations in 3 different sequences
Arm/Group | All Treated
Number analyzed (Participants) | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 30.7 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 10
  Black or African American | 2
  Asian | 0
  American Indian or Alaska native | 0
  Native Hawaiian or other Pacfic Islander | 0
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Median Scores on a Subjective Sweet Intensity Scale for Current and New Powder for Oral Use (POU) Formulations of Atazanavir
Description: Tasting atazanavir (15 mg, administered as a 5 mL oral suspension) was defined as taking the sample into the mouth, swishing it across the tongue for approximately 30 seconds without swallowing, and then spitting it out. Immediately after tasting each treatment, participants scored the treatments for sweetness using a subjective sweet intensity scoring system: 0=not sweet, 1=mildly sweet, 2=moderately sweet, 3=very sweet. Participants were permitted to select a whole or half score number (for example, 1.5) between the minimum score of 0 and the maximum score of 3.0. The higher the score, the greater the sweetness.
Time Frame: Study Day 1
Population: All participants who tasted at least 1 dose of atazanavir
Measure: Median (Full Range); unit: Units on a scale
Groups:
- Atazanavir, 15 mg/5 mL, With 10% Aspartame: Participants tasted atazanavir, 15 mg/5 mL, powder for oral use (POU) in the current formulation with 10% aspartame (Treatment A).
- Atazanavir, 15 mg/5 mL, With 4.2% Aspartame: Participants tasted atazanavir, 15 mg/5 mL, in the first new POU (POU1) with 4.2% aspartame (Treatment B)
- Atazanavir, 15 mg/5 mL, With 4.2% Aspartame + 0.53% Sucralose: Participants tasted atazanavir, 15 mg/5 mL, in the second new POU formulation (POU2) with 4.2% aspartame plus 0.53% sucralose (Treatment C)
Arm/Group | Atazanavir, 15 mg/5 mL, With 10% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame + 0.53% Sucralose
Number analyzed (Participants) | 12 | 12 | 12
Units on a scale | 1.5 [0.5 to 2.0] | 1.5 [0 to 2.0] | 1.0 [0 to 2.5]

2. Secondary Outcome: Median Palatability Score for Current and New Powder for Oral Use Formulations of Atazanavir
Description: Overall palatability was scored on a scale of 1 through 5, with 1 being least palatable and 5 being most palatable. Only whole score numbers were accepted.
Time Frame: Study Day 1
Population: All participants who tasted at least 1 dose of atazanavir
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Atazanavir, 15 mg/5 mL, With 10% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame + 0.53% Sucralose
Number analyzed (Participants) | 12 | 12 | 12
Units on a scale | 3 [2 to 4] | 3 [1 to 4] | 2 [1 to 5]

3. Secondary Outcome: Mean Palatability Score for Current and New Powder for Oral Use (POU) Formulations of Atazanavir
Description: as for outcome 2
Time Frame: Study Day 1
Population: All participants who tasted at least 1 dose of atazanavir
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Atazanavir, 15 mg/5 mL, With 4.2% Aspartame: Participants tasted received atazanavir, 15 mg/5 mL, in the first new POU (POU1) with 4.2% aspartame (Treatment B)
Arm/Group | Atazanavir, 15 mg/5 mL, With 10% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame + 0.53% Sucralose
Number analyzed (Participants) | 12 | 12 | 12
Units on a scale | 3.0 (0.85) | 2.8 (1.11) | 2.3 (1.07)

4. Primary Outcome: Mean Scores on a Subjective Sweet Intensity Scale for Current and New Powder for Oral Use (POU) Formulations of Atazanavir
Description: as for outcome 1
Time Frame: Study Day 1
Population: All participants who tasted at least 1 dose of atazanavir
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Atazanavir, 15 mg/5 mL, With 4.2% Aspartame+ 0.53% Sucralose: Participants tasted atazanavir, 15 mg/5 mL, in the second new POU formulation (POU2) with 4.2% aspartame plus 0.53% sucralose (Treatment C)
Arm/Group | Atazanavir, 15 mg/5 mL, With 10% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame+ 0.53% Sucralose
Number analyzed (Participants) | 12 | 12 | 12
Units on a scale | 1.3 (0.66) | 1.4 (0.70) | 1.0 (0.62)

5. Secondary Outcome: Number of Participants With Marked Abnormalities in Results of Clinical Laboratory Tests
Time Frame: Study Day 1
Population: All participants who tasted at least 1 dose of atazanavir. No postdose clinical laboratory assessments were conducted because no participants swallowed any treatment blends.
Arm/Group | Atazanavir, 15 mg/5 mL, With 10% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame + 0.53% Sucralose
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Abnormal Findings on Electrocardiograms
Time Frame: Study Day 1
Population: as for outcome 5
Arm/Group | Atazanavir, 15 mg/5 mL, With 10% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame + 0.53% Sucralose
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Who Died and With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Study Day 1
Population: All participants who tasted at least 1 dose of atazanavir
Measure: Number; unit: Participants
Arm/Group | Atazanavir, 15 mg/5 mL, With 10% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame + 0.53% Sucralose
Number analyzed (Participants) | 12 | 12 | 12
Participants
  Deaths | 0 | 0 | 0
  AEs | 0 | 0 | 0
  SAEs | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Relevant Changes in Vital Signs
Time Frame: Study Day 1
Population: as for outcome 5
Arm/Group | Atazanavir, 15 mg/5 mL, With 10% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame + 0.53% Sucralose
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Study Day 1
Description: This was a taste assessment study; no participants swallowed any study drug.
Arm/Group | Atazanavir, 15 mg/5 mL, With 10% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame | Atazanavir, 15 mg/5 mL, With 4.2% Aspartame + 0.53% Sucralose
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
This was a taste assessment only; participants did not swallow any treatment blends.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.